CLINICAL TRIAL: NCT05589844
Title: A Phase 1b Safety and Immunogenicity Study of Cytomegalovirus (CMV) Directed Type 1 Polarized Dendritic Cell Vaccination (αDC1) After Allogeneic Hematopoietic Cell Transplantation (alloHCT) for Hematologic Malignancies
Brief Title: A Cytomegalovirus-Directed Vaccine (CMV-alphaDC1) for Preventing Cytomegalovirus Infection or Reactivation in Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study never approved
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: I 1289721; NCI-2022-05780 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 1289721 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2022-10-17; First posted 2022-10-21 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Cytomegaloviral Infection; Hematopoietic and Lymphoid System Neoplasm
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Stem Cell Transplantation; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (CMV-alphaDC1) (Experimental): Patients undergo standard of care allogeneic hematopoietic stem cell transplant on day 0 and receive CMV-alphaDC1 vaccine intradermally on days 28, 42, 56, and 70.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Biological: CMV pp65 Peptide-loaded Alpha-type-1 Polarized Dendritic Cell Vaccine

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo standard of care allogeneic hematopoietic stem cell transplant
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Procedure: Biospecimen Collection — Correlative studies
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: CMV pp65 Peptide-loaded Alpha-type-1 Polarized Dendritic Cell Vaccine — Given intradermally
  Other Names: CMV pp65 Peptide-loaded Alpha-type-1 Polarized DC Vaccine; Cytomegalovirus pp65 Peptide Loaded Alpha-type 1 Polarized Dendritic Cell Vaccine

SUMMARY:
This phase Ib trial evaluates the safety and most effective dose of a cytomegalovirus (CMV) pp65 peptide-loaded alpha-type-1 polarized dendritic cell (CMV-alphaDC1) vaccination in patients who are undergoing an allogeneic hematopoietic stem cell transplant. CMV is an opportunistic infection that can occur or reactivate after allogeneic hematopoietic stem cell transplant as a result of immunosuppression. The CMV-alphaDC1 vaccine is made of white blood cells that have been exposed to molecules called cytokines, as well as CMV proteins. Introducing these dendritic cells to the patients immune system may activate an immune response to CMV, protecting against infection or reactivation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety of cytomegalovirus (CMV) pp65 peptide loaded alpha-type 1 polarized dendritic cell (CMV-alphaDC1) vaccination after allogeneic hematopoietic cell transplantation (alloHCT).

II. Determine the immunogenicity of CMV-alphaDC1 vaccination after alloHCT.

SECONDARY OBJECTIVES:

I. Evaluate the effect of CMV-alphaDC1 vaccination after alloHCT on late CMV reactivation.

II. Evaluate the effect of CMV-alphaDC1 vaccination after alloHCT on non-relapse mortality (NRM).

EXPLORATORY OBJECTIVES:

I. Assess the effect of CMV-alphaDC1 vaccination on T cell subsets. II. Assess the effect of CMV-alphaDC1 vaccination on T cell receptor diversity.

OUTLINE:

On day 0, patients undergo standard of care hematopoietic stem cell infusion. Patients receive CMV-alphaDC1 vaccine intradermally on days 28, 42, 56, and 70.

After completion of study treatment, patients are followed up at days 84, 100, 180, and 365.

ELIGIBILITY:
Inclusion Criteria:

* Recipient age >= 18 years of age
* The recipient is CMV seropositive
* The recipient is planned to receive an allogeneic peripheral blood stem cell graft
* The recipient is planned to receive fludarabine, melphalan, and total body irradiation for the transplant conditioning regimen
* The recipient is planned to receive micro-dose methotrexate, tacrolimus, and mycophenolate mofetil for acute graft versus host disease (GvHD) prophylaxis
* The recipient has an expected hematopoietic cell transplantation-comorbidity index (HCT-CI) score of 4 or less based upon the data available at the time of eligibility assessment
* The recipient must understand the investigational nature of this study and has signed an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedures
* The donor is CMV seronegative or seropositive
* The donor is 8/8 human leukocyte antigen (HLA) (DR-B1, A, B, C) matched to the recipient
* The donor is willing and able to donate peripheral blood mononuclear cells in addition to peripheral blood stem cells
* The donor is willing to sign informed consent

Exclusion Criteria:

* The recipient is CMV seronegative
* The recipient is planned to receive T cell depletion in vivo (anti-thymocyte globulin [ATG], alemtuzumab, post-transplant cyclophosphamide) or ex vivo (alpha-beta T cell depleted or CD34+ selected grafts) as acute GvHD prophylaxis
* The graft source is cord blood or bone marrow
* The donor or recipient has HLA DRB1*0301 or DRB1*1501 alleles
* The recipient has a very high disease risk index (DRI) based upon the data available at the time of eligibility assessment
* The recipient has a medical, behavioral, or social condition which in the opinion of the investigators would preclude compliance with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-11-16 (Estimated); Study Completion 2025-11-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities | Up to 2 years
  For each dose level of cytomegalovirus (CMV) pp65 peptide loaded alpha-type 1 polarized dendritic cell (CMV-alphaDC1) vaccination that is tested. Will be summarized by dose level using frequencies and relative frequencies.
Number of multifunctional CMV antigen specific T cells | At days 28 (before vaccination), 42 (before vaccination), 56, 70, 84, 100, 180, 365
  The number of multifunctional CMV antigen specific T cells will be determined by flow cytometry before and after vaccination with CMV-alphaDC1. Assessed by the change in the number of CMV specific T cells before and after treatment, which is compared using a one-sided paired t-test. The number of CMV specific T cells will be summarized before and after treatment using the appropriate descriptive statistics, with the mean change estimated using a 90% confidence interval.
Number of CMV pp56 reactive T cells | At days 28 (before vaccination), 42 (before vaccination), 56, 70, 84, 100, 180, 365
  The number of CMV pp65 reactive T cells will be determined by cytokine secretion (such as IFN-gamma) with ELISPOT before and after vaccination with CMV-alphaDC1. Assessed by the change in the number of CMV specific T cells before and after treatment, which is compared using a one-sided paired t-test. The number of CMV specific T cells will be summarized before and after treatment using the appropriate descriptive statistics, with the mean change estimated using a 90% confidence interval.

SECONDARY OUTCOMES:
Incidence of late CMV reactivation after allogeneic hematopoietic stem cell transplant | From day 85 to 365
  Will be summarized by dose level using the appropriate descriptive statistics; with estimates of rates obtained by 95% Jeffrey's prior confidence intervals.
Incidence of non-relapse mortality after allogeneic hematopoietic stem cell transplant | Up to 2 years
  Will be summarized by dose level using the appropriate descriptive statistics; with estimates of rates obtained by 95% Jeffrey's prior confidence intervals.

OTHER OUTCOMES:
Number of T cells | 1 year
  Includes CD4 T-cells, CD8 T-cells, delta gamma T-cells, and natural killer T-cells. Will be modeled as a function of time (treated as discrete) and random subject effect (through use of an auto-regressive covariance structure) with a linear mixed model. Mean differences of interest (i.e., changes after vaccination) will be evaluated by using Holm-Bonferroni adjusted tests on the appropriate contrasts of model estimates. All model assumptions will be evaluated graphically, and transformations will be applied as appropriate.
T cell receptor diversity | 1 year
  Measured by Vbeta spectra-typing. Will be modeled as a function of time (treated as discrete) and random subject effect (through use of an auto-regressive covariance structure) with a linear mixed model. Mean differences of interest (i.e., changes after vaccination) will be evaluated by using Holm-Bonferroni adjusted tests on the appropriate contrasts of model estimates. All model assumptions will be evaluated graphically, and transformations will be applied as appropriate.
Incidence of adverse events | Up to 2 years
  Toxicities and adverse events (as per Common Terminology Criteria for Adverse Events version 5.0) will be summarized by attribution and grade using frequencies and relative frequencies.

CONTACTS AND LOCATIONS:
Overall Officials: George L Chen, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States